CLINICAL TRIAL: NCT05830773
Title: Resonance Breathing Opioid Use Disorder
Brief Title: Resonance Breathing Intervention Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Fiona Conway, Assistant Professor, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000590
Record Dates: First submitted 2023-03-30; First posted 2023-04-26 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Substance-Related Disorders
Keywords: opioid use disorder; resonance breathing; substance use disorder; heart rate variability; drug craving
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: A convenience sample of participants are chosen for the intervention. There is no waitlist or control condition,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App Trial (Experimental): Use of the smartphone app
  Interventions: Other: Resonance Breathing Exercises

INTERVENTIONS:
Other: Resonance Breathing Exercises — This intervention uses the Camera Heart Rate Variability (CHRV) smartphone application, a resonance breathing app that is available for download to iPhones and Android devices. The CHRV app uses Photoplethysmography (PPG) technology to measure heart rate. PPG is a noninvasive technology that uses a light source (the phone's flashlight) and a photodetector (the phone's camera lens) at the surface of one's skin to measure the volumetric variations of blood circulation. The app also has a timer (to allow the participant to see how long they use the app in each session). The iPhone version of the app also has a breathing pacer (a bar that moves up and down to show the participant when to inhale and exhale). Participants are instructed to initiate a resonance breathing session for at least 5 minutes every day and whenever they experience cravings, feel like they are going to relapse, feel anxious or stressed, or just want to feel calm.

SUMMARY:
This study aims to assess the feasibility of an intervention for the management of craving, stress, anxiety, and depression among people who use opioids via a resonance breathing smartphone app.

DETAILED DESCRIPTION:
Most evidence-based treatments for substance use disorders (SUD) require face-to-face interactions with individuals who comprise a recovery support network. However, in the moment relapse occurs, people in recovery are often not in the presence of these trusted individuals. This project aims to address this issue by providing people in recovery with an application (app) that can be added to phones and other mobile devices to help them manage cravings, anxiety, and stress triggers at the specific moments they feel compelled to use. The connection between an individuals mind and body works in both directions. Psychological distress can cause psychosomatic symptoms in the body (e.g., stress is related to multiple chronic health conditions), but individuals can also use their bodies to affect psychology aspects (e.g., exercise can improve mood by releasing endorphins). A similar scientific theory is the foundation of controlled breathing interventions for anxiety, stress, and drug cravings. Psychological distress can disrupt the balance of our Autonomic Nervous System (which is responsible for our fight or flight response to threat), but breathing exercises can restore balance and decrease stress. The goal of this study is to test the feasibility, utility, and efficacy of an app that delivers controlled breathing exercises.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, participants need to be the legal age of majority (18 years of age or older), have the ability to read and speak in English, and have a history of alcohol or illicit drug use.

Exclusion Criteria:

Individuals with no access to a smartphone phone with a data plan, inability to provide consent and having suicidal thoughts or psychotic episodes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Average rating of participant satisfaction with the app as assessed by the Acceptability of Intervention Measure | 8 weeks
  The measure has 4 items on a scale from 1 (completely disagree) to 5 (completely agree). Higher scores are better outcomes. The citation for the measure is Weiner BJ, Lewis CC, Stanick C, et al. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci 2017; 12(1):108.
Average rating of participant assessment that the app is appropriate for managing cravings, stress, and anxiety as assessed by the Intervention Appropriateness Measure | 8 weeks
  The measure has 4 items on a scale from 1 (completely disagree) to 5 (completely agree). Higher scores are better outcomes. The citation for the measure is Weiner BJ, Lewis CC, Stanick C, et al. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci 2017; 12(1):108.
Average rating of participant assessment of whether the app was easy and practical to use as assessed by the Feasibility of Intervention Measure. | 8 weeks
  Feasibility entails participant assessment of whether the app was easy and practical to use. The measure has 4 items on a scale from 1 (completely disagree) to 5 (completely agree). Higher scores are better outcomes. The citation for the measure is Weiner BJ, Lewis CC, Stanick C, et al. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci 2017; 12(1):108.

SECONDARY OUTCOMES:
Average rating of participant assessment of their frequency of drug craving as assessed by the Aggregated Drug Craving Scale. | 8 weeks
  The measure has 5 items on a scale from 0 (Never - 0 times over the past month) to 6 (Nearly all of the time - more than 40 times or more than 6 times per day). Lower scores are better outcomes. The citation for the measure is: Costello MJ, Viel C, Li Y, Oshri A, MacKillop J. Psychometric validation of an adaptation of the Penn Alcohol Craving Scale to assess aggregated drug craving. J Subst Abuse Treat 2020; 119:108127.
Average rating of participant assessment of their frequency of experieincing stress as assessed by the Peceived Stress Scale. | 8 weeks
  The measure has 10 items on a scale from 0 (Never) to 4 (Very Often). Lower scores a better outcomes. The citation for the measure is: Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. Journal of health and social behavior. 1983 Dec 1:385-96.
Average rating of participant assessment of their frequency of experieincing anxiety as measured by the Beck Anxiety Inventory. | 8 weeks
  The measure has 21 items on a scale from 0 (Not at all) to 4 (Severely). Lower scores are better outcomes. The citation for the measure is: Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol 1988; 56(6):893-7.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Conway, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- Online, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared

REFERENCES:
- [Background] Vafaie N, Kober H. Association of Drug Cues and Craving With Drug Use and Relapse: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2022 Jul 1;79(7):641-650. doi: 10.1001/jamapsychiatry.2022.1240. PMID 35648415
- [Background] Kennedy AP, Epstein DH, Jobes ML, Agage D, Tyburski M, Phillips KA, Ali AA, Bari R, Hossain SM, Hovsepian K, Rahman MM, Ertin E, Kumar S, Preston KL. Continuous in-the-field measurement of heart rate: Correlates of drug use, craving, stress, and mood in polydrug users. Drug Alcohol Depend. 2015 Jun 1;151:159-66. doi: 10.1016/j.drugalcdep.2015.03.024. Epub 2015 Apr 7. PMID 25920802
- [Background] Price JL, Bates ME, Morgano J, Todaro S, Uhouse SG, Vaschillo E, Vaschillo B, Pawlak A, Buckman JF. Effects of arousal modulation via resonance breathing on craving and affect in women with substance use disorder. Addict Behav. 2022 Apr;127:107207. doi: 10.1016/j.addbeh.2021.107207. Epub 2021 Dec 17. PMID 34953433
- [Background] Brzozowski A, White RG, Mitchell IJ, Beech AR, Gillespie SM. A feasibility trial of an instructed breathing course in prison to improve emotion regulation in people with substance use difficulties. The Journal of Forensic Psychiatry & Psychology 2020; 32(2):308-25.
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Costello MJ, Viel C, Li Y, Oshri A, MacKillop J. Psychometric validation of an adaptation of the Penn Alcohol Craving Scale to assess aggregated drug craving. J Subst Abuse Treat. 2020 Dec;119:108127. doi: 10.1016/j.jsat.2020.108127. Epub 2020 Sep 16. PMID 33138922
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Derived] Conway FN, Kane H, Dorsainvil M, Kennedy P, Cance JD. Mobile resonance frequency breathing smartphone application to support recovery among people with opioid use disorder: Study protocol for feasibility study. PLoS One. 2024 Jan 31;19(1):e0296278. doi: 10.1371/journal.pone.0296278. eCollection 2024. PMID 38295049